CLINICAL TRIAL: NCT07251699
Title: COMBINED EFFECT OF EARLY WEIGHT BEARING AND ACTIVE KNEE EXERCISES IN TREATMENT OF TIBIAL PLATEAU FRACTURES WITH INTERNAL FIXATION
Brief Title: EFFECT OF EARLY WEIGHT BEARING AND ACTIVE KNEE EXERCISES IN TREATMENT OF TIBIAL PLATEAU FRACTURES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohmed yehia elabd hasan, phyisical therapist at qena oncology center, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tibial plateau early rehab
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Tibial Plateau Fractures
Keywords: early reabilitation
MeSH Terms: conditions — Tibial Plateau Fractures

STUDY DESIGN:
Intervention Model Description: A triple-blinded clinical randomized trial: (the research assistant, the participants, and the statistician) will be blinded to the treatment groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A triple-blinded clinical randomized trial: (the research assistant, the participants, and the statistician) will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A will receive early active knee ROM exercises with weight 24 bearing. (Experimental): Group A
  Early active exercises will be applied from the first day by the participation of the patient with the assistance of the physiotherapist as follows:
  Weeks: 1-4
  The program will be applied according to (Mohamed et al., 2022) as follows:
  Week: 1
  Day: 1-2:
  1. Static quadriceps, hamstrings and glutei.
  2. Static abdominal and back exercises.
  3. Active knee flexion and extension ROM exercises as possible according to patient tolerance and pain.
  Day: 3-4:
  In addition to the previous we add the following
  1. Ankle toe movement.
  2. Active exercises of the unaffected limb.
  3. Respiratory exercises. 33
  4. Cryotherapy.
  5. Active assisted hip abduction (0° -10°).
  6. Ankle toe movement; heel slides (0°-5°). Day: 5-7
  In addition to previous exercises, the following exercises will be added:
  1. Half bridging exercise.
  2. Active SLR (0°-15°).
  3. Active abduction (0°-15°).
  4. Active adduction (15°-0°).
  5. Heel slides (0°-10°). Weight bering excecises Ten percent of load on the affect leg
  Interventions: Other: Early active exercises will be applied from the first day by the participation of the patient with the assistance of the physiotherapist
- Group B will receive early passive ROM with delayed weight bearing. (Active Comparator): Passive ROM will be applied from the first day according to (Arslan, A et al., 2015) and late weight bearing based on (Amin et al.,2023) as follows:
  Weeks: 1-4
  1. Cryotherapy for 10 minutes three times per day.
  2. Passive exercises:
     1. ROM exercises.
     2. Passive ankle toe movements for 10 repetitions.
     3. Passive knee flexion as tolerated The program will be applied without active participation from the patient. It will be applied by the physiotherapist.
  3. Weight bearing is mainly in the sound side not affected so no weight bearing in the affected limb for about four weeks (Amin et al., 2023).
  Weeks: 5-8 Same protocol as Group A. Weeks: 9-12 Same protocol as Group A. Weeks: 13-16 Same protocol as Group A. The difference between each group is in the first four weeks and the type of program group one started with active exercise from the first day 38 group 2 active exercises started from week five at the first four weeks program is done by passive ROM modalities and by the physiotherapis
  Interventions: Other: Early active exercises will be applied from the first day by the participation of the patient with the assistance of the physiotherapist

INTERVENTIONS:
Other: Early active exercises will be applied from the first day by the participation of the patient with the assistance of the physiotherapist — The difference between each group is in the first four weeks and the type of program group one started with active exercise from the first day 38 group 2 active exercises started from week five at the first four weeks program is done by passive ROM modalities and by the physiotherapist. Early weight bearing is early in group 1 from the first week and late in group 2 after four weeks

SUMMARY:
This study will answer the following research questions:

Are there any significant differences between combination of early active knee ROM exercises and weight bearing versus early passive ROM with delayed weight bearing on pain intensity, ROM knee flexion and extension, function, and radiological healing in treatment of patients with TPFs fixed with plates and screws?

DETAILED DESCRIPTION:
This study will be conducted to compare the effects of combining early active knee ROM exercises and weight bearing versus early passive ROM and delayed weight bearing on pain intensity, ROM knee flexion and extension, function, and radiological healing in treatment of patients with TPFs fixed with plates and screws.

Tibial plateau fractures are associated with unfavorable outcomes due to a variety of factors, including soft tissue envelopes and cartilage damage, comorbidities such as compartment syndrome, postoperative infection, stiffness or malfunction of the knee, and even post-traumatic osteoarthritis (Narang et al., 2021). Consequently, they not only present surgical challenges but also have serious negative effects on function and quality of life (Arnold et al., 2017; Bhamra and Naqvi, 2021).

Physical therapy including active exercises is well supported in literature but in the late phases of rehabilitation. The concept of introducing early active exercises to patients undergoing rehabilitation following TPFs repaired with implants isn't well-supported in the literature. There aren't any comprehensive studies that specifically examine the application of early active exercises for TPFs repaired with plates and screws (Phansopkar et al., 2022).

There are few studies in form of case reports that applied early active exercises for patients with TPFs. It was found that appropriate surgical intervention followed with planned exercise protocol focussing on long term benefits can greatly help patients with TPFs to achieve early pain free mobility in lower limbs (Narang et al., 2021; Arya and Harjpal, 2023; Bhure et al., 2022).

this study will assess the long term effects of the treatment program for patients with TPFs fixed with plates and screws. So this study will be conducted, using valid and reliable methods and instrumentations, to determine if there are any effects of combined effect of early active 6 exercises and early weight bearing in treatment of patients with TPFs fixed with plates and screws which will add a new step in the pyramid of evidence for the best treatment methods for patients with TPFs fixed with plates and screws.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria Participants will be included in the study if they had TPF type II Schatzker fixed with plate and screws. Their aged range from 18-50 years old while their BMI range from 18.5 to 29.9 kg/m2 (Mohamed et 25 al., 2019; Hoseini et al., 2022; Phansopkar et al., 2022). They are referred from an orthopedic surgeon immediately after the operation.

Exclusion Criteria Participants will be excluded from this study if they didn't fulfil the inclusion criteria or if they had one of the following. Other types of TPFs or methods of fixation, previous hip or lower extremity injury or surgery e.g. arthroplasty, systemic diseases e.g. diabetes, rheumatoid arthritis, pathological conditions of the lower extremities e.g. tumours, infections, leg deformity, cardiovascular disease such as hypertension, and neurological diseases.

Exclusion Criteria:

-

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | 5 min
  This scale will be used to measure pain intensity. It is a valid and reliable scale for pain intensity measurement, (
Modified Rasmussen Radiologic Score | 5 min
  This chart is valid measurement tool for assessing fracture healing

SECONDARY OUTCOMES:
Universal Goniometer | 5 min
  This tool will be used to measure ROM of knee flexion and extension. The goniometer is a 360° protractor with one axis that joins two arms; a stationary arm and a movable one around the fulcrum of the protractor, (Figure 6). It is a valid and reliable tool in measurement of knee ROM (Acar et al., 2024).
Arabic version of the Knee injury and Osteoarthritis Outcome Score (KOOS) | 5 min
  This scale will be used to assess function. The KOOS scale's creators demonstrated the scale has excellent internal consistency, test-retest reliability, construct validity. In addition, it has responsiveness to variations in bodily function (Torad, A et al., 2015). The KOOS-AR is a valid indicator of activity limitation brought on by musculoskeletal problems of the lower 27 extremities. It also has excellent internal consistency and test-retest reliability with relatively small measurement error, (Appendix II), (Almangoush,.,et al., 2013).

CONTACTS AND LOCATIONS:
Overall Officials: enas fawzy mohamed, phd, Principal Investigator — Enas.fawzy@pt.cu.edu.eg
Locations (1):
- faculty of physical therapy cairo university, Giza,, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided